CLINICAL TRIAL: NCT02288351
Title: Intestinal Remodeling And Reprogramming of Glucose Metabolism Following Laparoscopic Roux-en-Y Gastric Bypass
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI decided to withdraw the study. No patient interaction took place.
Sponsor: Duke University (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00054934
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Roux-en-Y gastric bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Biopsy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RYGB with mucosal abnormality on EGD (Other): Subjects with Type 2 Diabetes undergoing a Roux-en-Y Gastric Bypass with a diagnosis of gastritis, esophagitis, ulcer, or other mucosal abnormality discovered at routine preoperative upper endoscopy, requiring follow-up endoscopy in the post-operative period.
  Interventions: Other: Mix Nutrient Meal; Other: labs; Other: Biopsy; Other: Second Mix Nutrient Meal; Other: Second biopsy; Device: PET/CT

INTERVENTIONS:
Other: Mix Nutrient Meal — Before Surgery: Subjects will have a visit where they will have a mixed nutrient stimulation test. They will be asked to fast for 12 hours prior to this visit (except water). During the visit they will drink an 8 ounce mixed nutrient liquid meal in 5 minute intervals over 20 minutes. During this visit a catheter will be placed in a vein in their arm for blood sample collections. A total of 50 ml of blood will be collected, (10 ml before drinking the mixed nutrient drink, at 30 minutes, at 60 minutes, at 90 minutes and 120 minutes after the mixed nutrient drink).
Other: labs — Fasting Plasma Glucose (FPG) and insulin will be added to the standard pre-operative labs.
Other: Biopsy — Intra-operatively: Subjects will undergo a standard laparoscopic Roux-en-Y Gastric Bypass (RYGB). During the surgery a 2cm tissue sample of the Roux limb will be taken by the doctor and frozen.
Other: Second Mix Nutrient Meal — 2 months post-operatively a second mixed nutrient stimulation test will be performed following the same process used pre-operatively.
Other: Second biopsy — . Patients will also be scheduled to undergo a second upper endoscopy and a 2cm biopsy of the Roux limb will be taken by the doctor and frozen in liquid nitrogen.
Device: PET/CT — Lastly, subjects will have a positron emission tomography/computed tomography (PET/CT) scan with Fluorodeoxyglucose (FDG) to evaluate the glucose in the Roux limb after surgery.

SUMMARY:
The purpose of this study is to investigate small intestinal remodeling and reprogramming of glucose metabolism in patients with Type 2 Diabetes Mellitus (T2DM) who undergo laparoscopic Roux-en-Y Gastric Bypass (RYGB). Our specific goal is to determine if the gene and protein expression levels of GLUT-1 are up regulated in the Roux limb and whether this is a major mechanism for the remission of T2DM following RYGB.

The two aims of the study are: 1) to demonstrate that the basement membrane glucose transporter 1 (GLUT-1) is upregulated in the Roux limb following RYGB, and 2) to demonstrate that the upregulation of GLUT-1 is a major mechanism for the improvement in glycemic control observed in T2DM patients undergoing RYGB.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 2 Diabetes Mellitus
2. Age between 18 and 65 years of age
3. BMI > 35kg/m²
4. Diagnosis of gastritis, esophagitis, ulcer, or other mucosal abnormality discovered at routine preoperative upper endoscopy, requiring follow-up endoscopy in the post-operative period.

Exclusion Criteria:

1. Patients undergoing revision from another bariatric procedure to RYGB
2. Presence of a seizure disorder (GLUT-1 deficiency syndrome)
3. Use of Tricyclic antidepressants
4. Use of tobacco products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Elevated Glut-1 gene and protein expression levels | 2 months
  Gene and protein expression levels of GLUT-1 will be analyzed from the specimens obtained intra-operatively (baseline) and at 2 months post-operatively to determine if levels are significantly elevated above baseline. Quantitative real-time PCR and Western blot techniques will be utilized as described in C below.

SECONDARY OUTCOMES:
Glut-1 level change in fasting glucose | 2 months
  Change in GLUT-1 levels will be correlated with changes in fasting glucose, mixed meal stimulation test, and homeostasis model assessment (HOMA). Secondly, at 2 months post-operatively, whole-body positron emission tomography/computed tomography (PET/CT) scanning with Fluorodeoxyglucose (FDG) will be performed to evaluate glucose uptake and utilization in the Roux limb.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Omotosho, MD, Principal Investigator — Duke University